CLINICAL TRIAL: NCT00513149
Title: Validation of the Clinical Applicability of Various Platelet Function Assessments in High-Risk Atherothrombotic Patients Undergoing Percutaneous Coronary Angioplasty: Phase 4 Study
Brief Title: Platelet Function Assessment for Atherothrombotic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Tzung-Dau Wang, M.D., Ph.D., NTUH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200612040R
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Coronary Artery Disease
Keywords: angioplasty; clopidogrel; coronary artery disease; PFA
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- c6 (Active Comparator): Clopidogrel 600 mg loading
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 600 mg loading

SUMMARY:
Background-Despite the pivotal pathogenic role of platelets in atherothrombosis has been widely recognized, there is a striking lack of consensus regarding how to measure platelet function and how to monitor the effects of various antiplatelet drugs. In view of the fact that recurrent ischemic events occurred in 8.5% to 8.8% of patients treated with dual antiplatelet drugs and there is significant inter-individual variability in platelet reactivity, we believe that the importance of platelet function assessment and its clinical implication should not be overlooked.

DETAILED DESCRIPTION:
Methods and Expected Results-In this prospective follow-up study, we will assess the predictive power of different assays of platelet function (PFA-100, plasma levels of von Willebrand factor, P-selectin, soluble CD40 ligand, and myeloid-related protein-8/14, and ADP-induced P-selectin [CD62P] expression on platelets by flow cytometry) before and after high-dose (600 mg) clopidogrel loading, at 3-month follow-up, and at study end on the occurrence of major cardiovascular events (MACE)(death, myocardial infarction, stroke, and coronary revascularization). We will also evaluate the correlations between different assays of platelet function. Based on our previous pilot study which demonstrated that a significant association between collagen-ADP closure time measured by PFA-100 and the occurrence of major cardiovascular events in 130 patients undergoing coronary angioplasty followed up for 6 months, we plan to include 150-200 patients into the present study. The total inclusion period is estimated to be 1 year. Therefore, a total of 2 to 2.5 years will be needed to complete this study. In the first year, we will analyze (1) the correlations between various platelet parameters and coronary angiographic findings; (2) the correlations among different platelet function measurements; and (3) the responsiveness of CADP-CT on high-dose clopidogrel loading.

In the second year, we will (1) analyze the predictability of various platelet parameters, at different point of time (baseline, after clopidogrel loading, at study end), on the occurrence of MACE and (2) establish a risk-prediction schema for patients undergoing coronary angioplasty. A pre-defined threshold value for the collagen-epinephrine closure time is set at 190 s, since this value has been recommended by other investigators to differentiate the presence or absence of aspirin resistance. A pre-defined threshold value for the collagen-ADP closure time is set at 90 s, since we found in our pilot study that this value was associated with the best discriminating ability for identifying patients developing MACE. In the third year, genetic background determining the PFA-100 closure time and levels of plasma markers of platelet activation will be explored by analyzing the relationships between various SNP/haplotype patterns and values of different platelet function assessments.

Clinical Significance-The present study will be the first to explore the clinical role of platelet function assessment both at baseline, after high-dose clopidogrel loading, and at study end. It may give us great insights regarding how to treat high-risk patients adequately with antiplatelet agents.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease

Exclusion Criteria:

* History of bleeding diathesis
* History of drug or alcohol abuse or liver disease
* Abnormal prothrombin time
* Abnormal platelet count
* Serum creatinine >1.5 mg/dl.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-07; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
the occurrence of major cardiovascular events (MACE)(death, myocardial infarction, stroke, and clinically driven target lesion revascularization) | 1 year

SECONDARY OUTCOMES:
the correlations between various platelet parameters and coronary angiographic findings | 1 year
the correlations among different platelet function measurements | 1 year
the responsiveness of CADP-CT on high-dose clopidogrel loading | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Dau Wang, M.D.,Ph.D., Study Chair — National Taiwan University Hospital
Locations (1):
- Division of Cardiology, Department of Internal Medicine and Department of Medical Imaging, National Taiwan University Hospital, Taipei, Taiwan